CLINICAL TRIAL: NCT00895154
Title: A Rehabilitation Program in Children With Sickle Cell Disease and Cognitive Deficits: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Society of Hematology (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Allison King, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 653; K23HL079073 (NIH)
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell; Memory; Learning; Achievement
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Tutoring Group (Active Comparator): Participants will receive general tutoring in the subject of his/her choice.
  Interventions: Behavioral: General Tutoring
- Tutoring + Memory Training Group (Experimental): Participants will receive tutoring and memory training.
  Interventions: Behavioral: General Tutoring; Behavioral: Memory Training

INTERVENTIONS:
Behavioral: General Tutoring — Participants will be tutored for approximately 8-10 hours per month during the school year.
Behavioral: Memory Training — Participants will receive memory training for approximately 8-10 hours per month during the school year.
  Arms: Tutoring + Memory Training Group

SUMMARY:
The overall goal of this project is to determine the feasibility of conducting a cognitive intervention for children with sickle cell disease.

DETAILED DESCRIPTION:
The primary aims of this clinical trial are:

1. Determine the effectiveness of targeted learning and memory strategy remediation in students with sickle cell disease and cognitive deficits.
2. Determine if there is improvement in academic achievement after targeted memory strategy remediation.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease that is confirmed by hemoglobin analysis
* Has a brain magnetic resonance imaging (MRI) document reading by a neuroradiologist
* Cognitive deficits, which are defined by one standard deviation lower than the normal ranges of an age-based standard score in cognitive tests that are evaluated by a psychologist
* Must be a student who will remain in school for at least 2 years
* Must provide informed consent with assent in accordance with the institutional policies (institutional review board approval)

Exclusion Criteria:

* Known developmental delays (these participants are ineligible because their learning potential may be biased from a prior insult)
* Intelligent quotient is less than 50 (may have impaired learning potential)
* Aphasic (i.e., unable to produce intelligible speech)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2003-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison King, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Yerys BE, White DA, Salorio CF, McKinstry R, Moinuddin A, DeBaun M. Memory strategy training in children with cerebral infarcts related to sickle cell disease. J Pediatr Hematol Oncol. 2003 Jun;25(6):495-8. doi: 10.1097/00043426-200306000-00014. PMID 12794531
- [Result] King AA, White DA, McKinstry RC, Noetzel M, Debaun MR. A pilot randomized education rehabilitation trial is feasible in sickle cell and strokes. Neurology. 2007 Jun 5;68(23):2008-11. doi: 10.1212/01.wnl.0000264421.24415.16. PMID 17548550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants are patients of the Pediatric Division of Hematology at Washington University School of Medicine and St. Louis University School of Medicine. Participants will be recruited during regularly scheduled clinic visits.
Pre-assignment Details: 21 patients completed informed consent to participate in the study. 3 withdrew before the start of the study so they were never assigned to study arms.
Groups:
- Tutoring + Memory Training Group: Participants will receive tutoring and memory training.
  General Tutoring: Participants will be tutored for approximately 8-10 hours per month during the school year.
  Memory Training: Participants will receive memory training for approximately 8-10 hours per month during the school year. Specific memory training strategies used will include silent rehearsal training and semantic clustering training.
Period: Overall Study
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Started | 8 | 10
Follow Up | 7 | 8
Completed | 7 | 8
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 10 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 18
Full Scale IQ (FSIQ); Wechsler Abbreviated Scale of Intelligence (WASI) [Mean (Standard Deviation); unit: Scores on a scale] — Participants engage in 4 subtests: Block Design, Vocabulary, Similarities, and Matrix Reasoning. Participants receive a raw score on each of these 4 subtests. This raw score is converted to a T score using a score chart in the WASI manual. The T scores from all 4 subtests are summed together to obtain a Full Scale Sum of T Scores. This Full Scale Sum of T Scores is converted to a Full Scale IQ-4 Composite Score using a score chart published in the WASI manual. Higher scores indicate better intelligence. FSIQ-4 Range: 40-160. Average FSIQ-4 =100, standard deviation is +/- 15.
  Scores on a scale | 85.13 (11.74) | 84.2 (11.35) | 84.61 (11.12)
Verbal IQ (VIQ); Weschler Abbreviated Scale of Intelligence (WASI) [Mean (Standard Deviation); unit: scores on a scale] — The VIQ score is comprised from the Vocabulary and Similarities subtests of the WASI-4. The raw scores from these subtests are converted to T scores using score charts in the manual. The T scores are summed together for a Verbal Sum of T Scores. This score is converted to a Composite VIQ score using a score chart in the manual. Higher scores = better Verbal IQ. Range = 45-160. Average = 100; standard deviation +/- 15.
  scores on a scale | 86.13 (13.74) | 89 (12.40) | 87.72 (12.70)
Performance IQ (PIQ); Weschler Abbreviated Scale of Intelligence (WASI) [Mean (Standard Deviation); unit: scores on a scale] — The PIQ score is comprised from the Matrix Reasoning and Block Design subtests of the WASI-4. The raw scores from these subtests are converted to T scores using score charts in the manual. The T scores are summed together for a Performance Sum of T Scores. This score is converted to a Composite PIQ score using a score chart in the manual. Higher scores = better Performance IQ. Range = 45-160. Average = 100; standard deviation +/- 15.
  scores on a scale | 87.13 (10.23) | 81.50 (13.97) | 84.00 (12.44)
Letter Word Identification subtest T score of Woodcock Johnson Psycho-Educational Battery (WS-III) [Mean (Standard Deviation); unit: scores on a scale] — This sub-test measures a student's word identification skills. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
  scores on a scale | 45 (10.57) | 45.78 (7.93) | 45.41 (8.97)
Reading Fluency subtest T score of WJ-III [Mean (Standard Deviation); unit: scores on a scale] — This sub-test measures a student's ability to read simple sentences quickly. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
  scores on a scale | 38.60 (10.015) | 49.00 (7.165) | 44.67 (9.652)
Calculations subtest T score of WJ-III [Mean (Standard Deviation); unit: scores on a scale] — This sub-test measures a student's ability to perform paper and pencil math computations.A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
  scores on a scale | 42.43 (9.95) | 44.38 (14.62) | 43.47 (12.26)
Math Fluency subtest T score of WJ-III [Mean (Standard Deviation); unit: scores on a scale] — This sub-test measures a student's ability to solve simple addition, subtraction and multiplication facts quickly. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
  scores on a scale | 35 (5.62) | 38.88 (9.51) | 37.21 (8.05)
Spelling subtest T score of WJ-III [Mean (Standard Deviation); unit: scores on a scale] — This sub-test measures a student's ability to write orally presented words correctly. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
  scores on a scale | 46.50 (8.54) | 45.67 (12.58) | 46.06 (10.54)
California Verbal Learning Test-Children's Version (CVLT-C) Trials 1-5 Immediate Recall T score [Mean (Standard Deviation); unit: scores on a scale] — The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
  scores on a scale | 42.75 (7.50) | 44.60 (11.70) | 43.78 (9.83)
CVLT-C Trials 1-5 Semantic Clustering T score [Mean (Standard Deviation); unit: scores on a scale] — The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The CVLT-C consists of five learning trials of 15 words which can be organized into three semantic categories. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
  scores on a scale | 54.38 (9.43) | 49.00 (11.01) | 51.39 (10.40)
CVLT-C Trials 1-5 Short Delay Recall T score [Mean (Standard Deviation); unit: scores on a scale] — The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
  scores on a scale | 44.88 (12.43) | 44.40 (7.83) | 44.61 (9.81)
CVLT-C Trials 1-5 Long Delay Recall T-Score [Mean (Standard Deviation); unit: scores on a scale] — The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
  scores on a scale | 45.00 (11.90) | 44.00 (9.67) | 44.41 (10.30)
CVLT-C Trials 1-5 Recognition Discriminability T score [Mean (Standard Deviation); unit: scores on a scale] — The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
  scores on a scale | 42.86 (17.29) | 45 (11.73) | 44.06 (13.93)
Delis Kaplan Executive Function System (D-KEFS) Number/Letter Switching T score [Mean (Standard Deviation); unit: scores on a scale] — The D-KEFS allows for the assessment of executive functions. There are 9 stand alone tests that can be individually or group administered. The Number-Letter Switching condition of the Trails Making sub-test specifically assesses flexibility of thinking on a visual-motor sequencing task. A participant's raw score (# of items answered correctly) is converted to a T score using tables provided in the manual. Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
  scores on a scale | 24.25 (3.40) | 41.40 (17.02) | 33.78 (15.20)

OUTCOME MEASURES:

1. Primary Outcome: Full Scale IQ (FSIQ) (WASI)
Description: The WASI is a brief, reliable measure of intelligence. Participants engage in 4 subtests: Block Design, Vocabulary, Similarities, and Matrix Reasoning. Participants receive a raw score on each of these 4 subtests. This raw score is converted to a T score using a score chart in the WASI manual. The T scores from all 4 subtests are summed together to obtain a Full Scale Sum of T Scores. This Full Scale Sum of T Scores is converted to a Full Scale IQ-4 Composite Score using a score chart published in the WASI manual. Higher scores indicate better intelligence. FSIQ-4 Range: 40-160. Average FSIQ-4 =100, standard deviation is +/- 15.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 86.43 (11.94) | 88.0 (10.94)

2. Primary Outcome: Verbal IQ (PIQ) (WASI)
Description: The VIQ score is comprised from the Vocabulary and Similarities subtests of the WASI-4. The raw scores from these subtests are converted to T scores using score charts in the manual. The T scores are summed together for a Verbal Sum of T Scores. This score is converted to a Composite VIQ score using a score chart in the manual. Higher scores = better Verbal IQ. Range = 45-160. Average = 100; standard deviation +/- 15.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 87.86 (13.79) | 87.78 (12.41)

3. Primary Outcome: Performance IQ (PIQ) (WASI)
Description: The PIQ score is comprised from the Matrix Reasoning and Block Design subtests of the WASI-4. The raw scores from these subtests are converted to T scores using score charts in the manual. The T scores are summed together for a Performance Sum of T Scores. This score is converted to a Composite PIQ score using a score chart in the manual. Higher scores = better Performance IQ. Range = 45-160. Average = 100; standard deviation +/- 15.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 87.29 (11.25) | 90.44 (9.98)

4. Primary Outcome: Letter Word Identification T Score (WJ-III)
Description: This sub-test measures a student's word identification skills. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 42.14 (7.01) | 44.00 (6.63)

5. Primary Outcome: Reading Fluency T Score (WJ-III)
Description: This sub-test measures a student's ability to read simple sentences quickly. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 40.14 (5.49) | 40.44 (7.65)

6. Primary Outcome: Calculations T Score (WJ-III)
Description: This sub-test measures a student's ability to perform paper and pencil math computations.A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 36.86 (9.55) | 44.56 (10.19)

7. Primary Outcome: Math Fluency T Score (WJ-III)
Description: This sub-test measures a student's ability to solve simple addition, subtraction and multiplication facts quickly. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 34.29 (4.86) | 38.56 (12.26)

8. Primary Outcome: Spelling T Score (WJ-III)
Description: This sub-test measures a student's ability to write orally presented words correctly. A participant's raw score (# of items answered correctly) is converted to a T score using a program (Compuscore for the WJ III, Version 2.1). Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 43.29 (6.95) | 44.22 (9.43)

9. Primary Outcome: California Verbal Learning Test-Children's Version (CVLT-C) List A Trials 1-5 Immediate Recall T Score
Description: The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 42.14 (12.77) | 36.90 (10.51)

10. Primary Outcome: CVLT-C Trials 1-5 Semantic Clustering T Score
Description: The CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The CVLT-C consists of five learning trials of 15 words which can be organized into three semantic categories. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 50.71 (7.87) | 43.70 (13.05)

11. Primary Outcome: CVLT-C Trials 1-5 Short Delay Recall T Score
Description: as for outcome 9
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 39.29 (13.67) | 34.50 (13.42)

12. Primary Outcome: CVLT-C Trials 1-5 Long Delay Recall T Score
Description: as for outcome 9
Time Frame: T scores were obtained at baseline and again at follow-up (after partcipant completed 50 hours of tutoring)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 40.00 (15.81) | 36.40 (14.48)

13. Primary Outcome: CVLT-C Trials 1-5 Recognition Discriminability T Score
Description: TThe CVLT®-C measures multi-trial learning and long-term recall abilities for verbal information. The Raw scores from all trials (1-5) are summed to calculate a Total Raw Score for Trials 1-5. This Raw score is converted to a T score using the CVLT-II Comprehensive Scoring System (computer system). A higher T score indicates better performance. Range = 0-100. Average =50 with a standard deviation of =/- 10 points.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 42.86 (16.07) | 37.50 (16.71)

14. Primary Outcome: Delis Kaplan Executive Function System (D-KEFS) Number/Letter Switching T Score
Description: The D-KEFS allows for the assessment of executive functions. There are 9 stand alone tests that can be individually or group administered. The Number-Letter Switching condition of the Trails Making sub-test specifically assesses flexibility of thinking on a visual-motor sequencing task. A participant's raw score (# of items answered correctly) is converted to a T score using tables provided in the manual. Higher T scores = better performance. Range: 0-100. Average T score = 50; standard deviation =/- 10.
Time Frame: After >/= 50 hours of tutoring
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
Number analyzed (Participants) | 7 | 8
scores on a scale | 33.67 (13.37) | 37.00 (15.42)

ADVERSE EVENTS:
Arm/Group | General Tutoring Group | Tutoring + Memory Training Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes